CLINICAL TRIAL: NCT03508817
Title: Randomized Clinical Trial on Atropine 0.01% for the Control of Myopia in Omani Children
Brief Title: Atropine 0.01% Eye Drops in Myopia Study
Acronym: AIMS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sultan Qaboos University (Other)
Collaborators: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Anuradha Ganesh, Senior Consultant, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MREC 1473
Record Dates: First submitted 2018-04-15; First posted 2018-04-26 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Myopia, Progressive
Keywords: Atropine, myopia, children
MeSH Terms: conditions — Myopia, Degenerative; Myopia | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Intervention group: Optimal myopia correction with single vision glasses and topical atropine 0.01%, one drop at night time.
  Control group: Optimal myopia correction with single vision glasses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine Sulfate 0.01% Eye Drops Group (Experimental): Intervention group will receive atropine sulphate eye drops 0.01% once nightly for 2 years.
  Interventions: Drug: Atropine Sulfate 0.01% Eye Drops
- Control group (No Intervention): Control group will not receive any medication.

INTERVENTIONS:
Drug: Atropine Sulfate 0.01% Eye Drops — atropine eye drop in study eye once nightly for two years.
  Other Names: Atropine
  Arms: Atropine Sulfate 0.01% Eye Drops Group

SUMMARY:
Control of myopia progression has become an important goal because of concerns regarding significantly increased risks of retinal degeneration, retinal detachment, glaucoma and cataract associated with high myopia. It is also clear there prevalence of myopia in children and young adults is increasing all over the world. Several methods including use of progressive addition lenses, rigid gas-permeable contact lenses, and life-style modifications (increased outdoor activity) have reported to alter myopia progression with varying efficacy. In general they have yielded clinical results of marginal significance. Atropine sulphate eye drops has consistently been demonstrated to inhibit axial myopia progression in both humans and animal models. Yet it has not found widespread clinical application for myopia control due to ocular side-effects of cycloplegia and pupil dilation. Recently 0.01% atropine has been shown to be effective in arresting myopia progression without side-effects of cycloplegia and near vision impairment and pupil dilatation and increased light sensitivity. Almost all studies on atropine have been carried out on children of Chinese origin. Efficacy (concentration and dosing) and safety need to be established in the population of interest, before routine use can be recommended. We plan to evaluate the efficacy and safety of topical 0.01% atropine eye drops in slowing the progression of myopia and ocular axial elongation in Omani children. A total of 150 children of ages 6-16 years will be randomized to two groups. Intervention group will receive atropine 0.01% once daily in each eye for two years (Phase 1). Control group will not receive any medications. Follow up visits will be scheduled every three months in Phase 1. Subsequently, medication will be stopped and the study patients will be followed up every six months for one year (Phase 2). The progression of myopia (change in refractive error and axial length) will be compared in the two groups by objective methods.

DETAILED DESCRIPTION:
To assess the efficacy and safety of using 0.01% atropine eye drops in reducing the progression of myopia in Omani population.

Objectives:

* To compare the effect of 0.01% atropine eye drops on progression of myopic refractive error and axial length with that in the control group.
* To study the effect of 0.01% atropine eye drops on pupil dilatation
* To study the effect of 0.01% atropine eye drops on amplitude of accommodation
* To study the effect of 0.01% atropine eye drops on near visual acuity
* To study the effect of 0.01% atropine eye drops on glare, photophobia and contrast senstivity

Research Methodology

Study design: Randomized, interventional, clinical trial.

Study population: Omani population (6 to 15 years of age) with myopia ≥ 2.00 < 8.00 Diopters (D).

Recruitment of participants: (1) Patients attending the pediatric ophthalmology out-patient department in Sultan Qaboos University Hospital (SQUH). (2) Children from primary schools.

Material:

WAM-5500 (Grand Seiko auto refractor/keratometer) Advanced binocular kerato-refractometer: The machine measures refraction, corneal curvature, pupil size and accommodation IOL master: 500 (Carl Zeiss; Meditec Inc, Dublin, CA) - Anterior chamber depth, axial length Standard Ophthalmic examination equipment

Study groups:

Intervention group: Optimal myopia correction with single vision glasses and topical atropine 0.01%, one drop at night time.

Control group: Optimal myopia correction with single vision glasses

Procedure:

1. Examination at enrollment (Eligibility Assessment): All eligible and willing subjects will undergo standard orthoptic and ophthalmic examination by one of the study investigators including measurement of best corrected visual acuity (both distant and near), accommodation, intraocular pressure, keratometry, cycloplegic refraction (autorefractor), slit lamp examination, and dilated fundus examination. Axial length, pupil size, anterior chamber depth will be measured. Cycloplegic refraction will be done 45min after instillation of cyclopentolate 1.0% eye drop (one drop every three times in 5min intervals)
2. Written informed consent will be obtained from the parents or legal guardians after thorough explanation of the nature and risks of the study (with use of patient information leaflet) before enrollment.
3. Randomization: Subjects will be allocated to intervention or control group in a randomized manner. Block randomization will be done with the blocks of 6, 4 and 2 with 30%, 40% and 30% respectively. The randomization will be done using SAS 9.1 version software.
4. Allocation Concealment: The allocation of treatment based on the randomization will be done using opaque envelops. These envelops will be sealed. These envelopes will be organized in an ascending order and will be kept in a binder folder and the binder clips will be sealed. This folder will be handed over to the Pharmacy department at the SQUH. These will be prepared at the Statistics and Health Information Department at the SQUH.
5. Phase 1: Intervention: Intervention group will receive atropine sulphate 0.01% once nightly for 2 years. Control group will not receive any medication. Atropine 0.01% minims will be made available by Pharmacy at SQUH. To aid and monitor compliance with the treatment regimen, each child / care-giver will be given a small calendar to tick off the days when the eye drop is instilled.
6. Phase 2: 1 year follow up after cessation of atropine 0.01% eye drops
7. Examination at follow up:

Follow up visits will be scheduled at 2 weeks following enrollment - base line measurements. Phase 1: 3 monthly intervals. Phase 2: 6 monthly intervals thereafter.

All assessments will be performed by investigators. A study coordinator will assess i) compliance with medication by checking the calendar, and ii) presence of any drug related discomfort using a questionnaire. Subsequently measurement of best corrected visual acuity, accommodation, pupil size, intraocular pressure, cycloplegic refraction, accommodation, axial length, anterior chamber depth slitlamp examination and dilated fundus examination (6 monthly intervals) will be carried out.

Outcome measures:

Efficacy. The primary outcome was progression of myopia, defined as the change in spherical equivalent refractive error (SER) relative to baseline. The assessment at 2 weeks after commencement of treatment will be considered at baseline value. This is necessary because atropine induces an additional cycloplegic effect that could lower further the SER. As such, a run-in period allows stabilization of the cycloplegic effect, thus making comparison of SER between the baseline and subsequent visits more meaningful. The SER is computed at each follow up visit. The secondary outcome is change in axial length during follow-up relative to baseline measured by A-scan ultrasonography.

Safety. The primary safety outcome monitored will be the occurrence of adverse events. The adverse effects description from previous studies include pupil dilation, photophobia, loss of accommodation, near visual impairment, and allergic response. Patients / parents will be questioned regarding glare, photophobia, contrast sensitivity, or any other adverse effects (questionnaire). Response to adverse events - The relationship of the event to the study medication will be assessed by the investigators as none, unlikely, possible, or definite. If patients experience glare / photophobia due to pupillary dilatation, they will be advised photochromic spectacles. Near adds will be advised in case of problem with near vision. Atropine will be discontinued in case of allergic response to medication.

Placebo effect:

The control group in our study will not receive any medication. Myopia progression will be assessed by objective (automated) methods - i.e. use of autorefractor for measuring change in refractive error and use of IOL-Master for measuring axial length. Side effects from use of atropine will also be measured objectively by quantifying pupil size and accommodation. Since there is no scope for bias from either the patient or the examiner in the above assessments, we believe that administering placebo drops as tear substitute would add to the cost and study protocol without added benefit.

Study duration: 3years

Statistical methods:

1. Sample size calculation:- The mean (SD) of progression myopia in the control is 0.75D (0.25D). In order to expect 20% reduction in the progression in the atropine arm with 90% power and 5% alpha error with two sided test, we need to study 58 subjects in each arm. However, incorporating 30% drop out we need to study about 75 subjects in each arm.
2. Data management: The data will be entered and managed in EPIDATA software enables with quality control checks. Double data entry will be done by the research assistant who is blinded. Queries will be generated and sent to the investigator and the corrections received will be updated in the database with the approval of the Research Officer or PI of the project. The data will be imported to SPSS for further analyses.

4. Analysis of results:

1. Pre-analysis Statistical Review Basic frequencies and distribution tables and/or plots will be performed for each variable. For example, histograms will be made for continuous variables and bar graphs will be generated for categorical variables.
2. Analyses of the Primary Outcome:

   The primary outcome (change in myopia) will be analysed using Intention To Treat (ITT) principles. The mean difference of myopia progression between the two groups will be computed with 95% CI, if the outcome is continuous variable and follows Normal distribution. Otherwise, bootstrapping will be done to establish 95%CI for the difference between two groups in the outcome and Mann Whitney U test will be done to test the hypothesis.However, the primary outcome will be further evaluated using Per Protocol (PP) principle, by excluding the cases who have had Protocol deviations. Secondary outcome (change in axial length) will be analysed and reported appropriately.
3. Safety Analysis set (As Treated Analyses set):

A separate dataset will be established for Adverse Events (AE) . These AE will be analysed using non parametric tests.. The analysis for safety includes all subjects, according to the route of intervention that they received and with at least one safety assessment. In addition, we will summarize explicitly any severe reactions or serious adverse events (SAE) in subjects received the wrong allocation.

Timing of Analyses and Stopping rule:

Two interim analyses will be done. One at the end of 1 year and another at the end 2 years. The stopping rule will be based Pocock method for 2 interim analyses. That is p<0.01 level will be considered as significant during the interim analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 to 15 years
* Myopia ≥ 2.00 D (cycloplegic refraction; spherical equivalent)
* No prior or current treatment for preventing myopia progression (bifocals / progressive addition lenses / orthokeratology)

Exclusion Criteria:

* Best corrected visual acuity < 0.5 (6/12)
* Refractive Myopia
* Astigmatism ≥ 1.5 D
* Amblyopia
* Ocular hypertension / Glaucoma
* Prior intraocular surgery
* Allergy to atropine eye drops
* Systemic diseases associated with myopia such as Marfan syndrome, Stickler syndrome
* History of cardiac or significant respiratory diseases
* Lack of consent for participating in the study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is progression of myopia | 2 years
  defined as the change in spherical equivalent refractive error (SER) relative to baseline

SECONDARY OUTCOMES:
change in axial length | 2 years
  change in axial length during follow-up relative to baseline measured by A-scan ultrasonography

OTHER OUTCOMES:
monitor of adverse events | 3 years
  The adverse effects description from previous studies include pupil dilation, photophobia, loss of accommodation, near visual impairment, and allergic response.

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Ganesh, MD, Principal Investigator — Sultan Qaboos University
Locations (1):
- Sultan Qaboos University, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Gong Q, Janowski M, Luo M, Wei H, Chen B, Yang G, Liu L. Efficacy and Adverse Effects of Atropine in Childhood Myopia: A Meta-analysis. JAMA Ophthalmol. 2017 Jun 1;135(6):624-630. doi: 10.1001/jamaophthalmol.2017.1091. PMID 28494063